CLINICAL TRIAL: NCT04982250
Title: Peer PrEP Referral + HIV Self-test Delivery for PrEP Initiation Among Young Kenyan Women: Pilot Study & Randomized Trial
Brief Title: Peer PrEP Referral + HIV Self-test Delivery for PrEP Initiation in Kenya
Acronym: PeerPrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katrina Ortblad, Assistant Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RG1121770; K99MH121166 (NIH)
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: HIV Prevention
Keywords: Kenya; adolescent girls and young women (AGYW); HIV pre-exposure prophylaxis (PrEP) delivery; HIV self-testing delivery

STUDY DESIGN:
Intervention Model Description: The pilot study will be a single group model (anticipated N=104), and the RCT will be a parallel model (anticipated N=400).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Enhanced peer PrEP referral + HIVST delivery" (Experimental): After a brief training, young female PrEP users will be encouraged to refer up to 4 peers to PrEP using strategies gained from the training, PrEP educational materials (i.e., brochures), HIVST kits (2 kits/peer = 8 kits total), and Kenya MOH-style referral cards.
  Interventions: Behavioral: Enhanced peer PrEP referral + HIVST delivery
- "Standard peer PrEP referral" (No Intervention): Young female PrEP users will be encouraged to refer 4 peers to PrEP using informal word-of-mouth recruitment strategies and Kenya MOH-style referral cards.

INTERVENTIONS:
Behavioral: Enhanced peer PrEP referral + HIVST delivery — After a brief training, young female PrEP users will be encouraged to refer up to 4 peers to PrEP using strategies gained from the training, PrEP educational materials (i.e., brochures), HIVST kits (2 kits/peer = 8 kits total), and Kenya MOH-style referral cards.
  Arms: "Enhanced peer PrEP referral + HIVST delivery"

SUMMARY:
Few young women at risk of HIV infection are initiating pre-exposure prophylaxis (PrEP) for HIV prevention in Kenya, thus we propose refining and testing a new model to increase PrEP initiation among young women at high HIV risk that has never been explored: enhanced peer PrEP referral with HIV self-test (HIVST) delivery. We conducted formative research to design of a model that is acceptable to young women and feasible to implement in Kenya. In this study, we will refine this model where young (≥16 to 24 years) female PrEP users refer their peers to PrEP and deliver HIVSTs in a pilot study and then test the refined model in a hybrid effectiveness-implementation trial. We hypothesize that relative to standard informal word-of-month peer PrEP referral (currently ongoing in Kenya), enhanced peer PrEP referral with HIVST delivery will increase PrEP initiation, continuation, and adherence among peers; have high fidelity; and be low cost.

DETAILED DESCRIPTION:
HIV PrEP is highly effective, but uptake remains low among young women in Africa, one of the populations at greatest HIV risk. In Kenya, one of the target groups for HIV incidence reduction is young women (16-24 years), who account for 33% of the total of new HIV infections yet comprise only 10% of the population. Barriers to PrEP initiation for this population are multi-faceted and include institutional (e.g., stigma associated with use) and intra-personal (e.g., lack of PrEP knowledge or self-efficacy) barriers. Thus, innovative PrEP delivery models that can overcome these barriers are needed. The opinion of peers often influences the behaviors and preferences of young women, including those related to health and health care. Most young women who have initiated PrEP in Kenya to date have done so because of informal peer referral, thus peer referral enhanced with training and HIVST delivery has the potential to increase PrEP initiation among members of this population. HIVST is a new technology that has the potential to enhance peer PrEP referral. Much of the emphasis on HIVST to date has been on identifying new individuals living with HIV and facilitating linkage to treatment, but most individuals who self-test will test negative and may be interested in starting prevention services, like PrEP.

We hypothesize that an enhanced peer PrEP referral model with HIVST delivery can increase PrEP initiation among young Kenyan women at HIV risk compared to standard informal peer PrEP referral. We conducted formative qualitative research to inform the design of such a model and propose refining this model in a pilot study with 16 young female PrEP users (i.e., "peer providers" or "index peers") who will be encouraged to referred up to four peer (i.e., "peer clients" or "referred peers"; =64 in total) using the defined implementation strategies (i.e., formalized training on PrEP and HIVST, and HIVST delivery). At one month, we will measure model adoption (e.g., peer referral, PrEP initiation) and feasibility (e.g., peer follow up) using survey data and qualitatively measure model acceptability using focus group discussions (FDGs) with index and referred peers (4-5 FDGs, 3-6 women/FDG).

We will incorporate findings from the pilot into a refined version of the enhanced peer PrEP referral with HIVST delivery model and test this compared to standard peer PrEP referral in hybrid effectiveness-implementation cluster-randomized controlled trial (cRCT). In our cRCT, we will randomize 80 index peers to either: 1) enhanced peer PrEP referral, where they are encouraged to refer 4 peer (i.e., "referred peers") to PrEP using an educational brochure, HIVSTs (2/peer), and a MOH-style referral slip, or 2) standard peer PrEP referral, where they are encouraged to refer 4 peer clients to PrEP using word-of-mouth, as is ongoing in Kenya, and a MOH-style referral slip. All trial outcomes will be measured among referred peers, as reported by index peers, three months later. Effectiveness outcomes will include PrEP initiation [primary], PrEP continuation (any refilling), and recent HIV testing (past 3 months); self-reported PrEP adherence will be assessed among referred peers reached for follow-up. Implementation outcomes will include model acceptability, fidelity, and costs. The results from this cRCT will address one of the greatest challenges to PrEP scale-up today and inform an R01 proposal for a community-randomized trial and budget impact analysis.

ELIGIBILITY:
Inclusion Criteria:

For peer providers (qualitative data, pilot):

* Age ≥16 to 24 years*
* Female
* Have been on PrEP for a minimum of three months
* Good adherence to PrEP (i.e., self-report take PrEP all the time)
* Willing to disclose PrEP use to their peers
* Able to identify up to 4 peers at risk of HIV infection
* Willing to participate in training with study counselors on PrEP referral and HIVST use
* Willing to refer peers to PrEP and deliver HIVSTs
* Able and willing to provide written informed consent
* Per the discretion of the site investigator, no clear risks of social harm or inability otherwise to reasonably conduct HIVST at home in the context of PrEP delivery

For peer providers (cRCT):

* Age ≥16 to 24 years*
* Female
* Must have refilled or initiated PrEP (i.e., been dispensed PrEP)
* Not currently enrolled in an HIV study
* Able to identify up to 4 peers with recent self-reported behaviors associated with risk of HIV acquisition
* Willing to participate in training with study counselors on PrEP referral and HIVST use
* Willing to refer peers to PrEP and deliver HIVSTs
* Able and willing to provide written informed consent
* Willing to provide contact information for follow-up
* Willing to engage in all research activities including completion of questionnaires
* Per the discretion of the site investigator, no clear risks of social harm or inability otherwise to reasonably conduct HIVST at home in the context of PrEP delivery

For peer clients (pilot, RCT):

* Age ≥16 to 24 years*
* Female
* Referred by peer (i.e., a PrEP users) to initiate PrEP
* Able and willing to provide informed consent

  * NOTE: We will only enroll young women ≥16 to 17 years into the study if they are emancipated minors and thus able to legally provide consent for participation in research. Kenyan law acknowledges women ages 14 to 17 who have become pregnant as emancipated minors. The PHRD site/UW collaboration has successfully enrolled emancipated minors into a number of prior studies, including PrEP clinical trials. In addition, Kenya's national policy guidelines explicitly permit PrEP use in this age group.

Exclusion Criteria:

For peer providers (qualitative data, pilot):

* Age ≥16 or >24 years
* Male
* Have not used PrEP for a minimum of three months
* Not willing to disclose PrEP use to their peers
* Not able to identify up to 4 peers at risk of HIV infection
* Not willing to participate in training with study counselors on PrEP referral and HIVST use
* Not willing to refer peers to PrEP and deliver HIVSTs
* Not able and willing to provide written informed consent

For peer providers (cRCT):

* Age ≥16 or >24 years
* Male
* Have not used PrEP
* Currently enrolled in an HIV study
* Not able to identify up to 4 peers at risk of HIV infection
* Illiterate
* Not willing to participate in training with study counselors on PrEP referral and HIVST use
* Not willing to refer peers to PrEP and deliver HIVSTs
* Not able and willing to provide written informed consent

For peer clients (pilot, cRCT):

* Age ≥16 or >24 years
* Male
* Not referred by peer (i.e., a PrEP users) to initiate PrEP
* Not able and willing to provide written informed consent

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 211 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katrina F Ortblad, ScD, MPH, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Partners in Health and Research Development, Thika, Kenya

IPD SHARING:
Plan to Share IPD: Yes
All data (deidentified) used for primary, secondary, and other outcomes reported in the main manuscript along with a data dictionary.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: September 2025 (around the time of publication). No end date.
Access Criteria: Anyone who wishes to access the data.
URL: https://github.com/Peer-PrEP-trial-Hutch/Peer-PrEP-main-manuscript

REFERENCES:
- [Background] Wilson IB, Lee Y, Michaud J, Fowler FJ Jr, Rogers WH. Validation of a New Three-Item Self-Report Measure for Medication Adherence. AIDS Behav. 2016 Nov;20(11):2700-2708. doi: 10.1007/s10461-016-1406-x. PMID 27098408
- [Derived] Wairimu N, Malen RC, Reedy AM, Mogere P, Njeru I, Culquichicon C, McGowan M, Gao F, Baeten JM, Ngure K, Ortblad KF. Peer PrEP referral + HIV self-test delivery for PrEP initiation among young Kenyan women: study protocol for a hybrid cluster-randomized controlled trial. Trials. 2023 Nov 4;24(1):705. doi: 10.1186/s13063-023-07734-x. PMID 37925450

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To identify index peers for recruitment, we reviewed the records of public clinics and research programs delivering PrEP in the region and called adolescent girls and young women (AGYW) who met the study eligibility criteria. Referred peers were recruited by index peers, who were given instructions to only recruit peers between 16 to 24 years who they thought might benefit from PrEP.
Pre-assignment Details: In both the pilot and the 2-arm cRCT, index peers (k) referred their peers to HIV services (i.e., referred peers, n). At follow-up, index peers reported outcomes for all the referred peers (started). At follow up, some of the referred peers were also enrolled (completed). Thus, some outcomes are measured among index peers, referred peers who started (as reported by index peers), and referred peers who completed (as reported by referred peers). Enrollment totals reflect those who completed.
Groups:
- Pilot: Index Peers (k): Index peers who received formalized training on PrEP referral strategies and HIV self-testing.
- Pilot: Referred Peers (n): Referred peers who were referred to HIV services by index peers.
- cRCT: Enhanced Group; Index Peers (k): Index peers assigned to the enhanced peer referral group.
- cRCT: Standard Group; Index Peers (k): Index peers assigned to the standard peer referral group.
- cRCT: Enhanced Group; Referred Peers (n): Referred peers who were referred to HIV services by index peers in the enhanced peer referral group.
- cRCT: Standard Group; Referred Peers (n): Referred peers who were referred to HIV services by index peers in the standard peer referral group.
Period: Overall Study
Arm/Group | Pilot: Index Peers (k) | Pilot: Referred Peers (n) | cRCT: Enhanced Group; Index Peers (k) | cRCT: Standard Group; Index Peers (k) | cRCT: Enhanced Group; Referred Peers (n) | cRCT: Standard Group; Referred Peers (n)
Started (Individuals counted as having started the study include:1) index peers who enrolled and completed baseline, and 2) all referred peers who were referred to PrEP by an index peer. Index peers reported outcomes for all these referred peers at follow-up.) | 16 | 56 | 40 | 42 | 137 | 104
Completed (Individuals counted as having completed the study include: 1) index peers who completed follow-up, and 2) referred peers who were referred to PrEP by an index peer and were subsequently enrolled in the study and completed a follow-up survey. This group reflects the total study enrollment and all those for whom we have demographic information.) | 16 | 30 | 40 | 42 | 55 | 28
Not Completed | 0 | 26 | 0 | 0 | 82 | 76
Not completed — Lost to Follow-up | 0 | 26 | 0 | 0 | 72 | 69
Not completed — Not Eligible to Enroll | 0 | 0 | 0 | 0 | 10 | 7

BASELINE CHARACTERISTICS:
Population: Of the 395 participants we have information about, only 211 were directly enrolled in the study and provided demographic information. These enrolled participants include index peers (k) and the subset of referred peers (n) we were able to enroll and follow-up, corresponding to those who completed the study in each population group.
Groups:
- Pilot: Referred Peers (n): Referred peers recruited by index peers whom we were able to reach for follow-up (completed enrollment).
- cRCT: Enhanced Group; Referred Peers (n): Referred peers recruited by index peers in the enhanced peer referral group whom we were able to reach for follow-up (completed enrollment).
- cRCT: Standard Group; Referred Peers (n): Referred peers recruited by index peers in the standard peer referral group whom we were able to reach for follow-up (completed enrollment).
- Total: Total of all reporting groups
Arm/Group | Pilot: Index Peers (k) | Pilot: Referred Peers (n) | cRCT: Enhanced Group; Index Peers (k) | cRCT: Standard Group; Index Peers (k) | cRCT: Enhanced Group; Referred Peers (n) | cRCT: Standard Group; Referred Peers (n) | Total
Number analyzed (Participants) | 16 | 30 | 40 | 42 | 55 | 28 | 211
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23 [21 to 24] | 21 [19 to 22] | 22 [20 to 23] | 22 [21 to 24] | 22 [20 to 23] | 22 [20 to 23] | 22 [20 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 30 | 40 | 42 | 55 | 28 | 211
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 16 | 30 | 40 | 42 | 55 | 28 | 211
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: cRCT: PrEP Initiation
Description: Number of referred peers that initiated PrEP, among all referred peers, as reported by index peers.
Time Frame: 3 months
Population: Outcome only applies to cRCT referred peers.
Measure: Count of Participants; unit: Participants
Arm/Group | cRCT: Enhanced Group; Referred Peers (n) | cRCT: Standard Group; Referred Peers (n)
Number analyzed (Participants) | 137 | 104
Participants | 41 | 41
Statistical Analysis 1: Comparison: cRCT: Enhanced Group; Referred Peers (n) vs cRCT: Standard Group; Referred Peers (n); The sample size calculation was based on the primary PrEP initiation outcome at follow-up; 80 clusters (40 per study group) provided 80% power to detect a 17% difference in PrEP initiation between the enhanced (80%) and standard (63%) groups, assuming three referred peers per cluster (75% of those recommended), an intra-cluster correlation coefficient of 0.05, and an alpha level of 0.05; Test type: Superiority; Risk Difference (RD) = -6, 95% CI 2-sided [-26 to 11] — Risk differences (RD) with 95% confidence intervals (CI) were estimated using regression models with Gaussian distributions, identify links, study group fixed effects, and index peer random effects (to adjust for clustering)

2. Primary Outcome: Pilot: PrEP Initiation, as Reported by Index Peers
Description: Number of referred peers that initiated PrEP, among all eligible referred peers, as reported by index peers.
Time Frame: 1 month
Population: Outcome only applies to pilot referred peers. The denominator (n=55) excludes one referred peer reported as HIV-positive.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot: Referred Peers (n)
Number analyzed (Participants) | 55
Participants | 43

3. Primary Outcome: Pilot: PrEP Initiation, as Reported by Referred Peers
Description: Number of referred peers that initiated PrEP, among eligible referred peers who enrolled and completed follow-up, as reported by referred peers.
Time Frame: 1 month
Population: Outcome only applies to pilot referred peers who enrolled and completed follow-up. The denominator (n=26) excludes four referred peers who were already/currently using PrEP at the time of referral.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot: Referred Peers (n)
Number analyzed (Participants) | 26
Participants | 22

4. Secondary Outcome: Pilot: PrEP Referral
Description: Number of referred peers referred to PrEP, among all referred peers, as reported by index peers.
Time Frame: 1 month
Population: Outcome only applies to pilot referred peers.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot: Referred Peers (n)
Number analyzed (Participants) | 56
Participants | 56

5. Secondary Outcome: Pilot: HIVST Use
Description: Number of referred peers that used HIVST, among referred peers who enrolled and completed follow-up, as reported by referred peers.
Time Frame: 1 month
Population: Outcome only applies to pilot referred peers who enrolled and completed follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot: Referred Peers (n)
Number analyzed (Participants) | 30
Participants | 29

6. Secondary Outcome: cRCT: Recent HIV Testing
Description: Number of referred peers who tested for HIV (any form, including HIVST) since peer PrEP referral, among all referred peers, as reported by index peers.
Time Frame: 3 months
Population: Outcome only applies to cRCT referred peers.
Measure: Count of Participants; unit: Participants
Arm/Group | cRCT: Enhanced Group; Referred Peers (n) | cRCT: Standard Group; Referred Peers (n)
Number analyzed (Participants) | 137 | 104
Participants | 125 | 56
Statistical Analysis 1: Comparison: cRCT: Enhanced Group; Referred Peers (n) vs cRCT: Standard Group; Referred Peers (n); Test type: Superiority; Risk Difference (RD) = 39, 95% CI 2-sided [24 to 54]

7. Secondary Outcome: cRCT: PrEP Continuation (Referred Peers)
Description: Number of referred peers that returned to a clinic to refill PrEP since referral, among all referred peers, as reported by index peers.
Time Frame: 3 months
Population: Outcome only applies to cRCT referred peers.
Measure: Count of Participants; unit: Participants
Arm/Group | cRCT: Enhanced Group; Referred Peers (n) | cRCT: Standard Group; Referred Peers (n)
Number analyzed (Participants) | 137 | 104
Participants | 17 | 11
Statistical Analysis 1: Comparison: cRCT: Enhanced Group; Referred Peers (n) vs cRCT: Standard Group; Referred Peers (n); Test type: Superiority; Risk Difference (RD) = 1, 95% CI 2-sided [-10 to 13]

8. Secondary Outcome: cRCT: PrEP Continuation (Index Peers)
Description: Number of index peers that returned to a clinic to refill PrEP in the past 3 months.
Time Frame: 3 months
Population: Outcome only applies to cRCT index peers.
Measure: Count of Participants; unit: Participants
Arm/Group | cRCT: Enhanced Group; Index Peers (k) | cRCT: Standard Group; Index Peers (k)
Number analyzed (Participants) | 40 | 42
Participants | 19 | 28
Statistical Analysis 1: Comparison: cRCT: Enhanced Group; Index Peers (k) vs cRCT: Standard Group; Index Peers (k); Test type: Superiority; Risk Difference (RD) = -19, 95% CI 2-sided [-40 to 2]

9. Secondary Outcome: cRCT: PrEP Adherence
Description: A 0-100 point PrEP adherence score derived from the validated three-item Wilson et al Adherence scale with higher scores indicating higher adherence, among referred peers who enrolled and completed follow-up, as reported by referred peers.
Time Frame: 3 months
Population: Outcome only applies to cRCT referred peers who enrolled and completed follow-up.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | cRCT: Enhanced Group; Referred Peers (n) | cRCT: Standard Group; Referred Peers (n)
Number analyzed (Participants) | 55 | 28
Scores on a scale | 4.9 [0.0 to 100.0] | 58.9 [0.0 to 100.0]
Statistical Analysis 1: Comparison: cRCT: Enhanced Group; Referred Peers (n) vs cRCT: Standard Group; Referred Peers (n); Test type: Superiority; Median Difference (Final Values) = -16.9, 95% CI 2-sided [-36.3 to 2.5]

10. Other Pre Specified Outcome: cRCT: PrEP Referral
Description: Median number of referred peers referred to PrEP services by each index peer.
Time Frame: 3 months
Population: Outcome only applies to cRCT index peers.
Measure: Median (Inter-Quartile Range); unit: referred peers
Arm/Group | cRCT: Enhanced Group; Index Peers (k) | cRCT: Standard Group; Index Peers (k)
Number analyzed (Participants) | 40 | 42
referred peers | 4.0 [3.0 to 4.0] | 3.0 [3.0 to 4.0]
Statistical Analysis 1: Comparison: cRCT: Enhanced Group; Index Peers (k) vs cRCT: Standard Group; Index Peers (k); Test type: Superiority; Median Difference (Final Values) = 0.5, 95% CI 2-sided [-0.2 to 1.1]

11. Other Pre Specified Outcome: cRCT: HIVST Use
Description: Number of referred peers in the enhanced group that used HIVST, among referred peers in the enhanced group who enrolled and completed follow-up, as reported by referred peers in the enhanced group.
Time Frame: 3 months
Population: We do not include the arm/group "cRCT: Standard group; referred peers (n)" here because this outcome only applies to referred peers in the enhanced group. Referred peers in the standard group did not receive HIVST as part of the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | cRCT: Enhanced Group; Referred Peers (n)
Number analyzed (Participants) | 55
Participants | 54

12. Other Pre Specified Outcome: cRCT: Linkage to Care
Description: Number of referred peers that went to a clinic to access HIV prevention or treatment services, among referred peers who enrolled and completed follow-up, as reported by referred peers.
Time Frame: 3 months
Population: Outcome only applies to cRCT referred peers who enrolled and completed follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | cRCT: Enhanced Group; Referred Peers (n) | cRCT: Standard Group; Referred Peers (n)
Number analyzed (Participants) | 55 | 28
Participants | 17 | 17

13. Other Pre Specified Outcome: cRCT: Materials Received
Description: Number of referred peers that received the intervention or standard-of-care materials, among referred peers who enrolled and completed follow-up, as reported by referred peers.
Time Frame: 3 months
Population: Outcome only applies to cRCT referred peers who enrolled and completed follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | cRCT: Enhanced Group; Referred Peers (n) | cRCT: Standard Group; Referred Peers (n)
Number analyzed (Participants) | 55 | 28
Participants | 46 | 24

14. Other Pre Specified Outcome: cRCT: Acceptability of Intervention Model
Description: Number of referred peers and index peers who agree/strongly agree (on a 5-point Likert scale) to statements adapted from the Theoretical Framework of Acceptability.
Time Frame: 3 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: cRCT: Appropriateness of Intervention Model
Description: Number of referred peers and index peers who agree/strongly agree (on a 5-point Likert scale) to statements adapted from the Appropriateness of Intervention Measure instrument.
Time Frame: 3 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: cRCT: Feasibility of Intervention Model
Description: Normal of referred peers and index peers who agree/strongly agree (on a 5-point Likert scale) to statements adapted from the Feasibility of Intervention Measure instrument.
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for index peers at both baseline and the month 3 follow-up visit, and for referred peers at the month 3 visit (so only collected among referred peers who enrolled and completed follow-up). During data collection and study follow-up, participants were asked to report if they've had any of these events and whether they are or are not study related.
Description: Adverse events (AEs) include any forms of verbal (e.g., yelling, fighting), physical (e.g., hitting), emotional (e.g., depression) or economic (e.g., job loss) abuse attributable to the study. While serious adverse events (SAEs) include hospitalization (for any condition, including those outside the study) or death.
Arm/Group | Pilot: Index Peers (k) | Pilot: Referred Peers (n) | cRCT: Enhanced Group; Index Peers (k) | cRCT: Standard Group; Index Peers (k) | cRCT: Enhanced Group; Referred Peers (n) | cRCT: Standard Group; Referred Peers (n)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/30 | 0/40 | 0/42 | 0/55 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/30 | 0/40 | 0/42 | 0/55 | 0/28
Other Adverse Events (participants affected / at risk) | 0/16 | 0/30 | 1/40 | 1/42 | 0/55 | 0/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pilot: Index Peers (k) (N=16) | Pilot: Referred Peers (n) (N=30) | cRCT: Enhanced Group; Index Peers (k) (N=40) | cRCT: Standard Group; Index Peers (k) (N=42) | cRCT: Enhanced Group; Referred Peers (n) (N=55) | cRCT: Standard Group; Referred Peers (n) (N=28)
Social Harms (Social circumstances) | 0 | 0 | 1 | 1 | 0 | 0 — Social harms include verbal (e.g., yelling, fighting), physical (e.g., hitting), emotional (e.g., depression) or economic (e.g., job loss) abuse attributable to the study.

LIMITATIONS AND CAVEATS:
Limitations included relying on index peers to report outcomes for referred peers in our primary analysis; low enrollment and follow-up among referred peers; relying on self-report for HIV testing and PrEP outcomes; and the relatively short follow-up period for all study participants (one month for pilot and three months for cRCT).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-06-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT04982250/Prot_002.pdf
  • Statistical Analysis Plan (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT04982250/SAP_003.pdf
  • Informed Consent Form (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT04982250/ICF_000.pdf